CLINICAL TRIAL: NCT06484296
Title: Training on Good and Green Health Practices in Midwifery Students Awareness Raising and Development of Good Health Practices Awareness Scale
Brief Title: Creating Awareness in Midwifery Students Through Training on Good and Green Health Practices and Awareness of Good Health Practices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Resmiye KAYA ODABAŞ, Asisstant Prof., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Resmiye-3
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Midwifery
Keywords: Mindfulness; Occupational Health Services; Climate Change
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Active Comparator): Before the training, students in all groups will be provided to take the Pretest.
  The students included in the training group will be trained on good and green health practices in the conference hall of the Faculty by expert researchers and the green transformation coordinator of the university who have a certificate of Conscious Awareness training. Three weeks after the training, all students will be given the Green Culture Scale Post-Test.
  Interventions: Other: Education
- Control Group (No Intervention): No application will be made to the control group. The students in this group will only fill in the questionnaires as pre-test and post-test three weeks after the pre-test.

INTERVENTIONS:
Other: Education — Before the training, students in all groups will be provided to take the Pretest.
  The students included in the training group will be trained on good and green health practices in the conference hall of the Faculty by expert researchers and the green transformation coordinator of the university who have a certificate of Conscious Awareness training. Three weeks after the training, all students will be given the Green Culture Scale Post-Test.
  Arms: Education Group

SUMMARY:
In this context, this study aims to increase midwifery students' awareness of good and green health practices and to develop a measurement tool to evaluate their awareness of good health practices. This research is in two stages, the first stage is methodological type, and the second stage will be carried out as a pre-test post-test randomized controlled experimental research between September 2024-2025. In the first stage, the Good Health Practices Awareness Scale will be developed. In the second stage of the study, the Green Culture Scale (pre-test-post-test) will be filled in by the students. The population of this study, which will be carried out in the Midwifery Department of Çanakkale Onsekiz Mart University, Faculty of Health Sciences, will consist of 300 students studying in the 2nd, 3rd and 4th grades of the Midwifery Department of this university. Data of the research; It will be collected with the "Introductory Information Form, Green Culture Scale and Good Health Practices Awareness Scale". Before starting to collect data, an item pool of the Good Health Practices Awareness Scale will be created in line with the literature, the measurement method will be determined and sent to at least ten faculty members who are interested in the subject and experts in the field, their opinions will be taken and scale items will be created in line with their opinions. Then, the purpose of the research will be explained to the students by the researchers and the groups the students belong to will be determined. Before the training, students in all groups will be asked to take the Pretest. Students included in the training group will be trained in good and green health practices in the faculty's conference hall by expert researchers with Conscious Awareness training certificates and the university's green transformation coordinator. Three weeks after the training, all students will take the Green Culture Scale Post-Test. Students in the control group will also receive training at an appropriate time. IBM SPSS Statistics 29 package program will be used for statistical analysis. In evaluating the data obtained as a result of the research, percentage rates, arithmetic mean and standard deviation, t test in dependent and independent groups and Bonferroni analysis will be used to determine where the significance comes from. Results will be evaluated at the 95% confidence interval and significance level of p < .05.

DETAILED DESCRIPTION:
Type (Design) of Research This research has two stages, the first stage is methodological type and the second stage will be carried out as a pre-test post-test randomised controlled experimental research. In the first stage, Good Health Practices Awareness Scale will be developed. In the second stage of the study, training will be given to Midwifery Department students about Good and Green Health Practices and the effectiveness of the training will be evaluated.

Population and Sample of the Study The research is planned to be conducted at Çanakkale Onsekiz Mart University, Faculty of Health Sciences, Department of Midwifery. The population of the study consists of 300 students studying in the 2nd, 3rd and 4th grades of the midwifery department of this university (based on the number of students in the 1st (n = 110), 2nd (n = 96) and 3rd (n = 94) grades of the 2023-2024 academic year). No sample selection will be made in the study, and it is planned that all 2nd, 3rd and 4th grade students will participate in the study. In scale studies, it is stated that the sample size should be at least ten times the number of items. Accordingly, the number of participants will be determined by multiplying the number of items in the scale by 10 to calculate the sample size. If the number of items determined is more than 30, first grade students will also be included in the study. For the second phase of the study, the students will be asked to participate in the training and control group (Training group: 150; Control group: 150). At the end of the research, the relevant sample size will be checked by post hoc power analysis. In the course curriculum of the Midwifery Department of this university, there is no course on environmental awareness, good practices, green practices, etc. In this respect, the variables that may affect the results of the study were tried to be taken under control.

Randomisation Full randomisation technique will be used to assign the participants to the groups. In the study, Random Lists website (https://www.randomlists.com/) was used and each class was divided into two groups by creating a random numbers table (n=150 for the education group and n=150 for the control group).

Data Collection Tools In the study, the data were collected using the "Descriptive Information Form, Green Culture Scale (GCS) and Good Health Practices Awareness Scale (GHPAS).

Introductory Information Form This form, created by the researchers in line with the literature (Perleth et al., 2001; Erötken & Durkan, 2010; Altındiş et al., 2018; Karasu, 2019), consists of two sections and a total of nine questions.

Green Culture Scale The adaptation study of the Green Culture Scale developed by Ermolaeva (2010), which will be used in the study, into Turkish was conducted by Ayyıldız Durhan et al. (2022). With the measurement tool obtained, it was aimed to examine the green culture levels of university students. 11 items and 2 sub-dimensions (Environmental Awareness and Environmental Behaviour), the total internal reliability coefficient was determined as 0.73. Within the scope of the two-stage study, the psychometric properties of the measurement tool were tested with 400 participants. Confirmatory factor analysis showed that the structure was confirmed. The validated structure shows that the original scale is suitable for use in the Turkish population. The increase in the score of the GAS, which was determined to be a valid and reliable measurement tool, indicates that the green culture level of the participants is high.

Good Health Practices Awareness Scale Before starting data collection, the item pool of the Good Health Practices Awareness Scale, which was created in line with the literature, was analysed during the scale development process.

will be created in accordance with the steps.

Data Collection and Training Process

Pre-Test Application After determining a suitable date for the training, the students in the training group completed the Introductory Information Form, Green Culture Scale (pre-test) before the training.

and Good Health Practices Awareness Scale. In the week when the training will be given, the students in the control group will be at school The participants will be asked to complete the Introductory Information Form, Green Culture Scale (pre-test) and Good Health Practices Awareness Scale in one day. Also, control The students in the group will be asked not to participate in the training and the students will be informed so that there is no interaction between the students.

Implementation of the Training Students studying in the Midwifery Department of the University and included in the training group will be given a training consisting of three sessions (with three lecturers) and lasting approximately three hours in total in the conference hall of the faculty at a time when their course programmes are suitable.

Final Test Application Three weeks after the training, students will be informed and asked to fill in the Green Culture Scale for the post-test without disrupting the class. Care will be taken not to disrupt the lesson. According to the literature, in order to evaluate the effectiveness of the training, it should be retested at least two weeks after the end of the training, ideally this period can be spread over three to six months, and up to one year for longer interventions.

Training the Control Group After the completion of the research, Good and Green Health Practices training will be given to the control group in order to avoid differences between the students without disrupting the education and training process. The date for the delivery of this training will be suitable for educators and students.

Data Evaluation

IBM SPSS Statistics 29 (Statistical Package for Social Sciences) package programme will be used for statistical analyses. Percentage ratios, arithmetic mean and standard deviation, t test in dependent and independent groups and Bonferroni analysis will be used to determine the source of significance. The results will be evaluated at 95% confidence interval and significance at p < .05 level. During the preparation of the scale, content validity analyses and construct validity analyses or factor analyses of a test used to measure a characteristic that cannot be measured directly will be performed during the creation of the scale items for expert acceptance.

ELIGIBILITY:
Inclusion Criteria:

* The participants were Çanakkale Onsekiz Mart University Midwifery Department 2nd, 3rd and 4th year students,
* Active students who attend the courses,
* Students who are willing and volunteer to participate in the study will be included.

Exclusion Criteria:

* Disabled to participate in the research,
* Has a diagnosed psychiatric diagnosis,
* Has a communication barrier,
* Students who do not continue their education and training (registration freeze) will be excluded from the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Awareness of Good and Green Health Practices | 3 weeks
  It will be applied as a pre-test together with the Good Health Practices Awareness Scale in order to determine the awareness levels of the students. Three weeks after the training, the same scale will be applied again as a post-test. The higher the score of the students, the better their awareness level will be understood.
Environmental Awareness and Environmental Behaviour | 3 weeks
  In order to determine the awareness levels of the students, it will be applied as a pre-test together with the Green Culture Scale. Three weeks after the training, the same scale will be applied again as a post-test. The higher the score of the students, the better their awareness level will be understood.

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye Demir, Ass. Prof, Study Director — Çanakkale Onsekiz Mart University; Resmiye Kaya Odabaş, Ass. Prof, Study Chair — Kocaeli University; Sibel Ocak Aktürk, Ass. Prof, Study Chair — Çanakkale Onsekiz Mart University; Neriman Güdücü, Ass. Prof, Study Chair — Kırklareli University